CLINICAL TRIAL: NCT01923077
Title: Early Intensive Treatment With Statins Improves Left Ventricular Function in Patients With Acute Myocardial Infarction.
Brief Title: Intensive Statin Therapy in Patients With AMI
Acronym: INTENSIFY
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Svendborg Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Soren Auscher, MD, ph.d-student., Svendborg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INTENSIFY
Record Dates: First submitted 2013-08-09; First posted 2013-08-14 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Acute Myocardial Infarction
Keywords: acute myocardial infarction; Statin; speckle tracking echocardiography; Strain; MSCT; plaque; vulnerable plaque
MeSH Terms: conditions — Sprains and Strains; Plaque, Amyloid | interventions — Simvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional (Placebo Comparator): Conventional treatment with simvastatin
  Interventions: Drug: Simvastatin
- Rosuvastatin (Active Comparator): loading dose of rosuvastatin 80 mg at randomization followed by 40 mg daily in 12 month.
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Simvastatin — usual care with Simvastatin
  Other Names: Simva
  Arms: Conventional
Drug: Rosuvastatin — rosuvastatin 80 mg as loading dose at randomization followed by rosuvastatin 40 mg daily.
  Other Names: crestor
  Arms: Rosuvastatin

SUMMARY:
Objective: Statins have been shown to have beneficial pleiotropic effects besides being lipid lowering. The investigators hypothesized that early and intensive statin treatment was associated with improved left ventricular (LV) function and with a stabilization of the coronary atherosclerotic plaques in patients with acute myocardial infarction (AMI) Method: In a prospective randomized blinded endpoint trial patients with ST segment elevation or non ST segment elevation AMI were randomized to either intensive statin-therapy (loading dose rosuvastatin 80 mg immediately after randomization followed by 40 mg daily) or usual statin therapy (simvastatin 40 mg daily). Patients were followed 12 month and the investigators performed echocardiography at randomization, after 30 days and after 12 month. The investigators used 2D Speckle Tracking for the assessment of LV-function. Coronary plaque assessment was done with Cardiac-CT (MSCT) at baseline and after 12 month.

Primary outcome for this study was assessment of LV function with global and regional myocardial strain. Secondary outcomes can be divided in 4 groups:

1. Additional echocardiographic measurements such as Ejection Fraction, S´, LV-volume, atrial volume, VA-coupling, diastolic function, post systolic strain and strain rate.
2. Biochemical assessment of inflammation and endothelial function: Hs-CRP, ICAM, VCAM, E-selection and Nitrate/Nitrite ratio.
3. Coronary plaque assessment by MSCT: Plaque volume and plaque stability.
4. Long term follow-up: Mortality and cardiovascular events

DETAILED DESCRIPTION:
Introduction Coronary heart disease (CHD) remains the leading cause of mortality in the western world. In Europe, CHD accounts for one fifth of all deaths annually. Acute myocardial infarction (AMI) is caused primarily by plaque rupture and it has been demonstrated that the pathogenesis of AMI involves interplay of the endothelium, the inflammatory cells and the thrombogenicity of the blood. Following an acute myocardial infarction (AMI), profound structural changes can be encountered, resulting in left ventricular (LV) remodeling and development of depressed cardiac function.

Heart failure (HF) is a significant cause of morbidity and mortality worldwide with an estimated prevalence of 1% to 2% in the western world and AMI remains the predominant cause.

Statins were first developed to improve the lipid profile and reduce the development of CVD. Several large randomized controlled trials have shown that statin therapy is beneficial in both primary and secondary prevention of atherothrombosis. Results from two large, acute coronary syndrome trials suggested further clinical benefit of statins in addition to their lipid lowering effect. This stemmed from the observation of a cardiovascular event-rate reduction in patients with AMI only weeks after initiation of statin treatment. Several experimental studies have demonstrated that statins, apart from their LDL lowering effect, exert beneficial pleiotropic effects on inflammation, endothelial function, thrombosis, plaque stability and ischaemic-reperfusion injury.Other experimental studies in animals have reported beneficial effects of statins on LV function after AMI. In clinical settings statins have been shown to prevent periprocedural myocardial damage in patients treated with percutaneous coronary intervention (PCI) and the ARMYDA-ACS trial demonstrated a protective effect of statin loading on the myocardium before PCI in patients with ACS. Only a few clinical studies have directly investigated the acute effect of statins on LV function in patients with AMI and the results are inconclusive.

All previous studies have concentrated on patients with STEMI and disregarded those with NSTEMI; moreover, no studies have investigated the effect of an early statin loading dose in patients with AMI. The investigators hypothesized that early and intensive statin treatment was associated with improved left ventricular (LV) function and with a stabilization of the coronary atherosclerotic plaques in patients with acute myocardial infarction (AMI) Thus, the primary aim of the Intensify trial was to examine the effect of early intensive statin treatment on LV function with strain echocardiography in patients with AMI after 30 days.

Methods Study population This study was a prospective randomized controlled (RCT) trial with a blinded endpoint design. The trial was approved by the Regional Scientific Ethics Committee for Southern Denmark and the Danish Data Protection Agency. Patients with AMI defined by current guidelines were consecutively collected from a single coronary care unit from April 2010-august 2012. Inclusion criteria were all patients with NSTEMI and STEMI, and the exclusion criteria were prior intensive statin treatment, contraindication to intensive statin therapy and a time limit above 24 hours from hospital admission.

Patients were randomized to either intensive statin treatment with rosuvastatin 40 mg or usual care with simvastatin 40 mg. The intensive care group was given a loading dose of rosuvastatin 80 mg as soon as possible followed by 40 mg daily. The usual care group was treated with simvastatin 40 mg daily. Apart from the different statin treatment, all patients were treated the same according to current national guidelines.

Patients were followed for 12 month and examined immediately after randomization, after 1 month and after 12 month.

Coronary angiography and Culprit vessel Culprit vessel and infarct location was identified from the coronary angiography. In patients with single vessel disease (lumen stenosis < 50%) the diseased vessel was identified as culprit. In patients with multi-vessel disease, the culprit vessel was identified by a combination of angiographic and electrocardiographic criteria. In patients with normal CAG we used electrocardiographic and multi-slice computer tomography to identify the culprit lesion. If the culprit lesion could not be found, the patient was excluded from the study. The investigators used the AHA scientific statement of myocardial segmentation and nomenclature for tomographic imaging from 2002 to define the coronary arteries supply area of the myocardium.

Echocardiography Echocardiography was performed at randomization and after 30 days using the GE Vivid 7 ultrasound system (GE Medical System Inc., Horten, Norway) with a standard 3.5 MHz ultrasound probe. A standardized protocol was followed at each examination and all examinations were performed by one operator. Consecutive heartbeats were recorded at a sweep speed of 25 mm/s and digitally stored, blinded to patient identity. Examinations were analyzed off-line by one experienced observer using EchoPAC version 1.12.0 (GE, Vingmed). All analysis was done with a sweep speed of 67 mm/s and recordings were measured and averaged from 3 consecutive heartbeats. Examinations with poor image quality and patients with atrial fibrillation were excluded from the analyses. Left ventricular- and atrial volumes were estimated using the Simpsons biplane method of discs in the 4- and 2 chamber views and ejection fraction was calculated. Mitral inflow pattern was estimated in the apical four chamber view and pattern of peak early (E) and peak atrial (A) velocities were measured. E/A ratio was calculated by dividing E by A. Mitral annular velocities were estimated in the apical 4- and 2 chamber view using pulsed wave tissue Doppler imaging. A pulsed wave Doppler sample volume was placed at the level of the mitral annulus first in the lateral wall, then in the septum and finally in the anterior- and posterior wall. Using tissue Doppler imaging peak early (E´), peak systolic (S´) mitral annular velocities were estimated. E/E´ ratio was obtained by dividing E by E´.

Strain analyses Longitudinal systolic strain was measured by speckle tracking echocardiography. This was obtained from 2D gray scale images of the apical 4-chamber, 2-chamber and long-axis view with optimized focus on the left ventricle and frame rate ≥ 69 frames/sec. Duration of systole was defined in the 5-chamber apical view by marking aorta valve opening and closure from the continuous wave Doppler curve.

Strain analyses were done in EchoPAC version 1.12.0 (GE, Vingmed) with the Q-analysis software. The left ventricular borderline was manually traced in each apical plane and tracking of motion was automatically done by the software. Peak systolic strain was determined in all 18 segments from the three apical views. Global strain for the left ventricle was provided by the software as the average value of the peak systolic longitudinal strain of the three apical views. Strain of the infarct zone was calculated as the mean value of the segments supplied by the culprit vessel

Time to intensive statin bolus:

Patients randomized to the intensive care group were given a loading bolus of rosuvastatin 80 mg as soon as possible after admission and continued intensive treatment with 40 mg daily. Patients randomized to the usual care group were treated after current guidelines with simvastatin 40 mg daily and started statin therapy before discharge from the hospital. Patients treated intensively were divided in two groups. A very early statin group receiving statin treatment before 12 hours after admission and an early statin group receiving statin after 12 hours but before 24 hours from admission to the hospital.

MSCT:

The investigators performed a contrast enhanced Cardiac CT (MSCT) at randomization and after 12 month. The investigators used a standardized protocol at every examination and detailed method description can be seen elsewhere.

Biochemistry:

Blood was drawn at baseline before randomization and after 30 days. The investigators measured lipid-profile HBA1C, Creatinin, ALAT and CK.

Statistical analyses Continuous outcome variables are presented as mean ± standard deviation (SD). Changes in outcome variables from baseline to follow-up are presented as Delta (∆) values (follow-up values - baseline values) Differences between groups are analyzed with an unpaired Students t-test with unequal variance. The investigators used multiple linear regressions in order to adjust for potential confounders. The investigators defined the confounders to be: Baseline left ventricular output variable, diabetes, hypertension, hypercholesterolemia, prior statin treatment, history of ACS, type of infarction, type of invasive treatment, culprit vessel, beta-blockers, ACE/ARB-inhibitors and time from symptoms to invasive treatment.

Continuous exposure variables are presented as median and lower and upper quartiles and categorical data as frequencies and percentages. Difference in exposure variables were tested with Krushal-Wallis test for continuous variables and for categorical variables with Fischer's exact test. Statistical tests were two-sided, and a P-value < 0.05 was considered to be statistically significant. All statistical analyses were performed using STATA version 12 (StataCorp LP, Collage Station, TX, USA)

ELIGIBILITY:
Inclusion Criteria:

* All patients with NSTEMI and STEMI

Exclusion Criteria:

* prior intensive statin treatment
* contraindication to intensive statin therapy
* Time limit above 24 hours from hospital admission.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-04; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Change in Global and Regional longitudinal systolic strain | baseline, 1 month and 12 month
  We want to investigate if early intensive statin treatment with rosuvastatin improve Global and Regional longitudinal systolic strain assessed by speckle tracking echocardiography compared to patients getting usual care with simvastatin 40 mg

SECONDARY OUTCOMES:
Change in LV-function assessed by 2D echocardiography: Ejection Fraction, S´, LV-volume, atrial-volume, VA-coupling, diastolic function. Post systolic strain(PSS) and strain rate | baseline, 1 month, 12 month
Change in endothelial function and inflammatory activity | baseline, 1 month and 12 month
  Endothelial function estimated by nitrate/nitrite ratio. Inflammatory response estimated by: hs-CRP, ICAM, VCAM, E-selectin,
Change in Coronary Plaque morphology | baseline and after 12 month
  Assessment of change in Plaque-volume and Plaque-morphology; Stabile Plaque vs. Vulnerable Plaque
Cardiovascular events and mortality | 5 years
  Follow-up after 5 years to register cardiovascular events and mortality

CONTACTS AND LOCATIONS:
Overall Officials: Søren SA Auscher, MD, Principal Investigator — OUH/Svendborg Hospital, Denmark
Locations (1):
- OUH/Svendborg Hospital, Svendborg, Funen, Denmark